CLINICAL TRIAL: NCT05660265
Title: A Randomized, Placebo-controlled, Double-Blind (Sponsor Unblind), Parallel Group, Single Dose, Dose Escalation Phase I Study in Sickle Cell Disease Participants, to Evaluate the Safety, Tolerability, and Pharmacokinetics of GSK4172239D
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Oral GSK4172239D Compared With Placebo in Sickle Cell Disease Participants Aged 18 to 50 Years
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study due to strategic business consideration and not related to safety.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 218471
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Diseases; Anaemia, Sickle Cell
Keywords: Hematologic diseases; Sickle cell disease; First time in human study; 218471
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: This is a placebo controlled multi-center study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be a double blinded study where the sponsor may be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Participants in this arm will receive either single dose of GSK4172239D (Dose 1) or matching placebo.
  Interventions: Drug: GSK4172239D; Other: Placebo
- Cohort 2 (Experimental): Participants in this arm will receive either single dose of GSK4172239D (Dose 2) or matching placebo.
  Interventions: Drug: GSK4172239D; Other: Placebo
- Cohort 3 (Experimental): Participants in this arm will receive either single dose of GSK4172239D (Dose 3) or matching placebo.
  Interventions: Drug: GSK4172239D; Other: Placebo
- Cohort 4 (Experimental): Participants in this arm will receive either single dose of GSK4172239D (Dose 4) or matching placebo.
  Interventions: Drug: GSK4172239D; Other: Placebo
- Cohort 5 (Experimental): Participants in this arm will receive either single dose of GSK4172239D (Dose 5) or matching placebo.
  Interventions: Drug: GSK4172239D; Other: Placebo
- Food effect cohort (Experimental): One selected cohort will also receive an additional single dose of GSK4172239D (or matching placebo) under fed (high calorie and high fat) conditions.
  Interventions: Drug: GSK4172239D; Other: Placebo

INTERVENTIONS:
Drug: GSK4172239D — Different strength of GSK4172239D will be administered in different cohorts.
Other: Placebo — Matching placebo will be administered.

SUMMARY:
This will be a first time in human (FTIH) study in sickle cell diseases (SCD) participants. The FTIH study is planned to evaluate the safety, tolerability, and pharmacokinetics of GSK4172239D.

The study will be composed of 3 periods for all participants (Screening, Treatment, and Follow up). Participants will be screened and, prior to first dose on Day 1, will be randomized to receive either GSK4172239D or placebo.

GSK4172239D is a prodrug that is converted in vivo into GSK4106401. This study will be a single dose, dose-escalation study. The initial dosing for all cohorts will be staggered so that 2 participants will be dosed as sentinel participants. Provided there are no safety concerns in 48 hours (h), the remaining 6 participants scheduled for the cohort may be dosed. One selected cohort of participants will also receive an additional single dose of GSK4172239D (or matching placebo) under fed (high calorie and high fat) conditions after a washout period of a minimum of 20 days or 5 half-lives, whichever is longer, designated as the Food Effect Cohort.

ELIGIBILITY:
Inclusion criteria:

* Participants diagnosed with SCD not taking medication which increases gamma-globin (fetal hemoglobin).
* Participants with SCD who have failed or not tolerated one or more approved therapies for SCD
* Body weight greater than (>) 50 kilogram (kg).
* For male participants: Refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR agree to use a male condom with female partner. Agree to use an additional highly effective contraceptive method with a failure rate of less than (<) 1% per year when having sexual intercourse with a woman of childbearing potential who is not currently pregnant
* For female participants: Female participants are eligible to participate if they are a woman of non-childbearing potential (WONCBP).
* Capable of giving informed consent.

Exclusion Criteria:

* Presence of active, clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data.
* Clinically significant abnormal blood pressure and/or history of hypertension as determined by the investigator.
* History of clinically significant heart disease as determined by the investigator.
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m^2
* ALT > 3x upper limit of normal (ULN).
* Bilirubin > 5x ULN (isolated bilirubin > 5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Hemoglobin < 6 gram/decalitre (g/dL).
* Absolute neutrophil count <1,500 / microlitre (μL).
* Platelet count <75,000 /μL or >750,000 /μL.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 t1/2 (whichever is longer) prior to the first dose of study drug, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise participant safety. By exception, participant may take acetaminophen (less than or equal to [≤] 2 g/day) up to 48h prior to the first dose of study drug.
* Use of hydroxyurea or decitabine within 9 weeks prior to baseline through follow-up.
* Blood transfusion within 3 months prior to baseline through follow-up.
* Current enrollment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study drug or any other type of medical research.
* Positive pre-study drug/alcohol screen. By exception, opioid use for pain or benzodiazepine use for anxiety as directed by a physician is permitted.
* Regular use of known drugs of abuse, except for use directed by a physician. By exception, opioid use for pain or benzodiazepine use for anxiety is permitted.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Area under curve zero to time infinity (AUC 0-inf) for GSK4106401 after a single oral dose of GSK4172239D | Up to Day 3
Maximum observed plasma concentration (Cmax) for GSK4106401 after a single oral dose of GSK4172239D | Up to Day 3
Time to Cmax (Tmax) for GSK4106401 after a single oral dose of GSK4172239D | Up to Day 3
Half-life (t1/2) for GSK4106401 after a single oral dose of GSK4172239D | Up to Day 3
Ratio between the fed and fasted conditions for AUC (0-inf) | Up to Day 3
Ratio between the fed and fasted conditions for Cmax | Up to Day 3

SECONDARY OUTCOMES:
Number of participants with clinically significant changes from baseline in white blood cell (WBC) | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in hemoglobin | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in platelets count | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in neutrophil count | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in alanine transaminase (ALT) | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in aspartate transaminase (AST) | Baseline and up to Day 7
Number of participants with clinically significant changes from baseline in bilirubin | Baseline and up to Day 7
Number of participants with adverse event (AE) and serious adverse event (SAE) | Up to Day 7
Number of participants with clinically significant change from baseline in 12 lead electrocardiograms (ECG) | Baseline and up to Day 7
Number of participants with clinically significant change from baseline in vital signs | Baseline and up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Riverdale, Georgia
  - GSK Investigational Site, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/